CLINICAL TRIAL: NCT02646202
Title: Scleroligation is a Safe and Effective New Technique for Eradication of Gastroesophageal Varices.
Brief Title: Scleroligation for Eradication of Gastroesophageal Varices.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Consultant liver and GIT diseases- Tanta university hospital, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scleroligation
Record Dates: First submitted 2016-01-01; First posted 2016-01-05 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Gastroesophageal Varices
MeSH Terms: interventions — Sclerotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sclerotherapy group (Active Comparator): thirty patients treated by sclerotherapy for OV using ethanolamine oleate 5%.
  Interventions: Procedure: Sclerotherapy
- Endoscopic band ligation group (Active Comparator): thirty patients treated by endoscopic banding using the Euro-Ligator system.
  Interventions: Procedure: Band ligation
- Sclero-ligation (SL) group (Experimental): thirty patients treated by intra variceal endoscopic sclerotherapy combined with band ligation.
  Interventions: Procedure: Scleroligation

INTERVENTIONS:
Procedure: Sclerotherapy — Injection of varices
  Arms: Sclerotherapy group
Procedure: Band ligation — endoscopic banding of varices
  Arms: Endoscopic band ligation group
Procedure: Scleroligation — intra variceal endoscopic sclerotherapy combined with band ligation.
  Arms: Sclero-ligation (SL) group

SUMMARY:
Gastric varices occur in 5-33% of patients with portal hypertension. Concomitant gastro esophageal varices are the most common type. Both endoscopic sclerotherapy and band ligation are very effective in controlling acute esophageal varices bleeding and preventing rebleeding.

DETAILED DESCRIPTION:
Evaluation of a new scleroligation technique for management of bleeding gastro-esophageal varices regarding efficacy, complications, variceal recurrence, and survival.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients presenting with an acute or recent episode of gastro-esophageal variceal bleeding.

Exclusion Criteria:

* Patients were excluded if they had malignancy of any origin.
* Any terminal illness, such as heart failure, uremia, or chronic pulmonary diseases.
* Other potential causes of GIT bleeding.
* Patients with previous endoscopic or surgical intervention for varices were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of sessions to complete variceal obliteration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ferial El-kalla, Professor, Principal Investigator — Head of endoscopy unit - Tropical medicine department- Tanta; Mohamed Elhendawy, Consultant, Principal Investigator — liver diseases dept.- Tanta university hospital; Loai Mansour, Consultant, Study Director — liver diseases dept.-Tanta university hospital; Abdelrahman kobtan, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Rehab Badawy, Consultant, Study Chair — liver diseases dept.-Tanta university hospital; Hanan Elbasat, Professor, Study Chair — liver diseases dept.-Tanta university hospital; Sherief Abd-Elsalam, Consultant, Study Chair — Liver diseases and gastroenterology dept.-Tanta university hospital
Locations (1):
- Tropical medicine dept.-Tanta university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mansour L, El-Kalla F, El-Bassat H, Abd-Elsalam S, El-Bedewy M, Kobtan A, Badawi R, Elhendawy M. Randomized controlled trial of scleroligation versus band ligation alone for eradication of gastroesophageal varices. Gastrointest Endosc. 2017 Aug;86(2):307-315. doi: 10.1016/j.gie.2016.12.026. Epub 2017 Jan 9. PMID 28082116